CLINICAL TRIAL: NCT07239531
Title: The Application of Interval Training in Advanced Life Support Skills Simulation Training for Medical Students: A Randomized Sequential Allocation Study
Brief Title: The Application of Intermittent Training in Clinical Skills Simulation Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Xinyu Zhan-2025-10
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Advanced Life Support Operational Skills and Theoretical Knowledge Learning and Memorization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval Training Group (Experimental): Conduct experiments on trainees who have mastered advanced life support theory and practical skills. The interval retraining group undergoes fixed-interval repeated training, performing the same 20-minute task daily on days 2, 4, and 6.
  Interventions: Other: Interval retraining
- Non-interval training group (Experimental): Conduct experiments on trainees who have mastered advanced life support theory and practical skills. Compared to the experimental group, this group of trainees will not receive additional training during the following week.
  Interventions: Other: Non-interval retraining

INTERVENTIONS:
Other: Interval retraining — Through basic skills training and testing, confirm that all trainees have mastered the steps of adult external cardiopulmonary resuscitation (CPR), tracheal intubation procedures, and the operational steps of automated external defibrillators (AEDs). And validated students' mastery of ECG interpretation for cardiac arrest and arrhythmias, along with pharmacology knowledge of cardiovascular emergency medications through assessment questions. The interval retraining group underwent fixed-interval repeated training, performing the same 20-minute tasks daily on days 2, 4, and 6.
  Arms: Interval Training Group
Other: Non-interval retraining — Through basic skills training and testing, confirm that all trainees have mastered the steps of adult external cardiopulmonary resuscitation (CPR), tracheal intubation procedures, and the operational steps of automated external defibrillators (AEDs). And validated students' mastery of ECG interpretation for cardiac arrest and arrhythmias, along with pharmacology knowledge of cardiovascular emergency medications through assessment questions. The non-interval retraining group will not engage in interval training during the following week.
  Arms: Non-interval training group

SUMMARY:
This study aims to investigate medical students' mastery of advanced life support skills when using scenario-based simulation combined with intermittent training, compared to traditional teaching methods.

DETAILED DESCRIPTION:
Advanced life support is crucial for medical students during their studies, examinations, and professional practice, serving as the foundation of their clinical skills. Scenario-based simulation training immerses students in realistic emergency scenarios, familiarizing them with equipment operation, fostering teamwork, and providing real-time feedback to mitigate clinical risks. Through scenario simulation, students encounter and manage authentic emergency situations within simulated clinical settings, thereby enhancing their skill proficiency and response capabilities. Intermittent training combined with deliberate practice helps medical students retain these skills and emergency knowledge over the long term. This study aims to investigate the impact of a teaching model integrating scenario simulation training with spaced practice, compared to traditional teaching methods, on medical students' long-term mastery of advanced life support theoretical knowledge and operational skills.

ELIGIBILITY:
Inclusion Criteria:

* Medical students studying in the Department of Anesthesiology
* The initial training for "Advanced Life Support Scenario Simulation Instruction" required by this study has been successfully completed, and the corresponding pre-test assessment has been passed.
* Voluntarily participate in this study and sign a written informed consent form, committing to adhere to the entire schedule of the research plan.
* During the research period, do not participate in any other training that conflicts with this experiment.

Exclusion Criteria:

* Individuals who have previously obtained an Advanced Cardiac Life Support (ACLS) provider certificate issued by the American Heart Association (AHA) or an equivalent organization, and whose certificate remains valid.
* Individuals who have participated in any form of Advanced Cardiac Life Support (ACLS) or Advanced CPR scenario simulation training courses within the past three months.
* Previously participated as a subject in educational interventions comparing "spaced learning versus traditional learning."
* Individuals who, for any reason, fail to complete all instructional components during the initial training phase or whose pre-test data is missing.
* Individuals who are unable to guarantee participation in all scheduled training or testing sessions during the study period (particularly on Days 2, 4, 6, and 7) due to scheduling conflicts, leave requests, or other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Advanced Life Support Skills Assessment | The seventh day after the unified training
  Performance Scoring for Cardiopulmonary Resuscitation, Defibrillation, and Tracheal Intubation
Theoretical Knowledge of Advanced Life Support | The seventh day after the unified training
  Interpretation of electrocardiograms related to cardiac arrest, arrhythmias, and other conditions; pharmacological knowledge of emergency medications for the cardiovascular system.

SECONDARY OUTCOMES:
Total Duration of Scenario Simulation | The seventh day after the unified training
  Total time required to resuscitate the patient in the simulated case
Scenario-Based Simulation Training Participant Behavior Checklist | The seventh day after the unified training
  Conduct standardized behavioral verification of trainees participating in scenario-based simulation training based on teaching cases.
Student Satisfaction Survey Form | The seventh day after the unified training
  Participant satisfaction with the training content and outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China